CLINICAL TRIAL: NCT05123118
Title: Lung and Breast Cancer Prevention by an Integrated Intervention of Maternal Smoking Cessation and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaozhong Wen (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Xiaozhong Wen, Associate Professor, State University of New York at Buffalo
Organization: State University of New York at Buffalo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00003067; UL1TR001412 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Smoking, Cigarette; Breastfeeding
Keywords: Pregnancy; Postpartum; Smoking abstinence; Breastfeeding intention; Breastfeeding duration
MeSH Terms: conditions — Cigarette Smoking; Breast Feeding | interventions — Lactation

STUDY DESIGN:
Intervention Model Description: The 40 eligible participants will be randomized into either the intervention (N=20) or control group (N=20). A sequence of random numbers in blocks of 2 will be used to ensure equal numbers of participants for each group over time.
Who Masked: Outcomes Assessor
Masking Description: Research staff who collect and analyze outcome data will be blinded to participants' group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated intervention (Experimental): Integrated intervention of smoking cessation and breastfeeding
  Interventions: Behavioral: Integrated intervention of smoking cessation and breastfeeding
- Attention placebo control group (Active Comparator): Instructions on general pregnancy and infant care
  Interventions: Behavioral: Attention placebo control

INTERVENTIONS:
Behavioral: Integrated intervention of smoking cessation and breastfeeding — The intervention group will receive an integrated intervention of smoking cessation and breastfeeding: education and counseling, monitoring and feedback, and contingent financial incentives.
  Arms: Integrated intervention
Behavioral: Attention placebo control — Participants in the control group will receive usual prenatal care from physicians, nurses, or social workers. They will receive best standard care on smoking cessation and breastfeeding, including referral to the New York State Smokers' Quitline and the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC).
  Arms: Attention placebo control group

SUMMARY:
This pilot clinical trial aims to integrate maternal smoking cessation and breastfeeding interventions to enhance both cancer prevention behaviors. The investigators will recruit 40 daily smoking women in their early pregnancy and randomize them into the integrated intervention or control group. Main outcomes include smoking abstinence and breastfeeding rates at 6 months postpartum.

DETAILED DESCRIPTION:
The investigators are proposing the first randomized controlled trial to integrate maternal smoking cessation and breastfeeding interventions to enhance both cancer prevention behaviors. The investigators will recruit 40 daily smoking women in their 1st or 2nd trimester of pregnancy (≤28 weeks) from local obstetric clinics, communities, and social media. They will be randomized into either the intervention (N=20) or control group (N=20). The two groups will complete the same number of sessions (6 during pregnancy and 3 postpartum), but focus on different topics. Specifically, the control group will receive instructions on general pregnancy and infant care. The intervention group will receive instructions on general pregnancy and infant care, plus an integrated multicomponent intervention that promotes both smoking cessation and breastfeeding (i.e., education and counseling, monitoring and feedback, and contingent financial incentives). Two female Certified Lactation Counselors (interventionists) will be trained to run study sessions during home visits. Interventionists will provide additional support via phone and text messaging until 6 months postpartum. Main outcomes include smoking abstinence and breastfeeding rates at 6 months postpartum within the duration of this award.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* At ≤28 weeks of pregnancy
* Daily smoking cigarettes and/or cigars in the past 7 days
* Be able to read, listen, and talk in English

Exclusion Criteria:

* Being diagnosed with cancer
* Current heavy drinking (more than 2 drinks a day)
* Current use of illicit substances
* Medical conditions contraindicating breastfeeding such as HIV infection, active tuberculosis, and breast removal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Wen, MD, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Division of Behavioral Medicine Department of Pediatrics Jacobs School of Medicine and Biomedical Sciences State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrated Intervention | Attention Placebo Control Group
Started | 20 | 20
Completed | 16 | 15
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Intervention | Attention Placebo Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 19 | 37
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Pregnancy status [Count of Participants; unit: Participants] — Pregnancy status is verified through testing the levels of human chorionic gonadotropin (hCG) in urine samples. If the urine hCG level is 20 mIU/mL or higher, the test shows a positive result, indicating pregnancy.
  Participants
    Pregnant | 20 | 20 | 40
    Not pregnant | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Abstinence
Description: Based on their recorded daily numbers of cigarettes and cigars smoked after enrollment, the investigators will classify smoking abstinence status in the past 7 days (7-day point-prevalence). The self-reported smoking abstinence will be biochemically confirmed by urine cotinine tests (<50 ng/mL).
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Intervention | Attention Placebo Control Group
Number analyzed (Participants) | 20 | 20
Participants | 8 | 3

2. Primary Outcome: Number of Participants With Reported Intent to Breastfeed
Description: During pregnancy, participants will report breastfeeding intention using questionnaires modified from the Infant Feeding Practices Study II. The question is, "What method do you plan to use to feed your new baby in the first few weeks?" with 4 response options: 1) breastfeeding only (baby will not be given formula), 2) formula feed only, 3) both breastfeed and formula feed, or 4) unsure. We create a binary variable to indicate breastfeeding intentions (option 1 or 3) or other feeding intentions (option 2 or 4).
Time Frame: 35 weeks of pregnancy (the end of pregnancy)
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Intervention | Attention Placebo Control Group
Number analyzed (Participants) | 20 | 20
Participants | 16 | 10

3. Primary Outcome: Number of Participants Reporting to Breastfeed
Description: During postpartum, mothers report their breastfeeding status (exclusive, mixed with formula, non-breastfeeding) every month until 6 months postpartum. Any breastfeeding is defined as exclusive breastfeeding or mixed-feeding breast milk and formula.
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Intervention | Attention Placebo Control Group
Number analyzed (Participants) | 16 | 15
Participants | 6 | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Integrated Intervention | Attention Placebo Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT05123118/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT05123118/ICF_001.pdf